CLINICAL TRIAL: NCT01563341
Title: Tandem DBS for Parkinson's Disease: A Pilot Study Utilizing STN/GPi + Hypothalamic Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ryan Uitti, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-007086
Record Dates: First submitted 2012-03-20; First posted 2012-03-26 (Estimated); Results first posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Parkinson's Disease; Deep Brain Stimulation
MeSH Terms: conditions — Parkinson Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Deep Brain Stimulation (Experimental): Parkinson's disease patients who would otherwise be undergoing subthalamic nucleus (STN) deep brain stimulation (DBS) will have dual hemispheric stimulation of the STN and globus pallidus interna (GPi).
  Interventions: Device: Deep brain stimulation

INTERVENTIONS:
Device: Deep brain stimulation — Study will be utilizing multiple brain electrodes simultaneously. The study will require at least two electrodes to be placed in one cerebral hemisphere (one for motor improvement and one for potential cognitive implications).

SUMMARY:
Does dual hemispheric stimulation of the subthalamic nucleus (STN) and fornix/hypothalamus potentially improve cognitive function in patients with Parkinsons disease.

ELIGIBILITY:
Inclusion Criteria:

* All patients will be enrolled from the practice of the primary investigator.
* Parkinson's Disease (PD) patients in whom optimal medical therapy has failed.
* All patients will have responsivity to levodopa.
* Individuals with normal or mild cognitive impairment.

Exclusion Criteria:

* Clinically significant dementia
* Other significant neurological or psychiatric disease
* Previous brain surgery including pallidotomy or thalamotomy
* Previous placement of other implantable devices

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-04; Primary Completion 2023-10-18 (Actual); Study Completion 2023-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Uitti, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Deep Brain Stimulation: Parkinson's disease patients who would otherwise be undergoing subthalamic nucleus (STN) deep brain stimulation (DBS) will have dual hemispheric stimulation of the STN and globus pallidus interna (GPi).
  Deep brain stimulation: Study will be utilizing multiple brain electrodes simultaneously. The study will require at least two electrodes to be placed in one cerebral hemisphere (one for motor improvement and one for potential cognitive implications).
  % participants were enrolled and underwent subthalamic nucleus (STN) deep brain stimulation (DBS) will have dual hemispheric stimulation of the STN and globus pallidus interna (GPi).
Period: Overall Study
Arm/Group | Deep Brain Stimulation
Started | 5
Completed | 0
Not Completed | 5

BASELINE CHARACTERISTICS:
Groups:
- Deep Brain Stimulation: Parkinson's disease subjects with dual hemispheric stimulation of the subthalamic nucleus (STN) and fornix/hypothalamus
Arm/Group | Deep Brain Stimulation
Number analyzed (Participants) | 5
Age, Customized [Mean (Full Range); unit: years] | 61.2 [55 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 5
Unified Parkinson's Disease Rating Scale [Median (Full Range); unit: units on a scale] — UPDRS was developed to evaluate various aspects of PD including non-motor and motor experiences of daily living and motor complications (total of 55 items). It includes a motor evaluation and characterizes the extent and burden of disease across various populations. Each item on the scale is rated as 0 being normal and 4 being severe. We only computed the motor section of the scale (29 items) Subjects scoring a total score of 0 would mean no symptoms and a score of 116 on the motor score would mean severe symptoms. The higher the sum of motor subsection (29 items) the worse the PD symptoms.
  units on a scale | 24 [0 to 116]

OUTCOME MEASURES:

1. Primary Outcome: Change in Memory Testing From Presurgical Baseline to 12 Months
Description: Memory will be assessed with the Hopkins Verbal Learning Test. The test consists of a set of six forms. Each test includes a list of 12 nouns; the examiner reads the list to the examinee, who repeats as many words as remembered. This process is repeated three times; 20-25 minutes later, examinees are asked again to recall as many words as possible; for the final task, the examiner reads a list of 24 words (including the 12 words from the list) and asks the examinee after each whether the word was on the list. For interpreting findings, in each metric listed on a scale from 0 to 12 with zero being worse and 12 being best (total recall, delayed recall, retention), higher scores reflect better learning efficiency (total recall) and memory (delayed recall, retention). Since this is a longitudinal study, follow-up scores will be compared to baseline. A positive direction of change would be interpreted as "improved" and a negative direction of change would be interpreted as "declined".
Time Frame: baseline, 12 months
Measure: Median (Full Range); unit: score on a scale
Groups:
- Deep Brain Stimulation: Parkinson's disease patients with dual hemispheric stimulation of the subthalamic nucleus (STN) and fornix/hypothalamus
Arm/Group | Deep Brain Stimulation
Number analyzed (Participants) | 4
score on a scale | 1 [0 to 5]

ADVERSE EVENTS:
Time Frame: Baseline to 12 Month
Description: Parkinson's disease subjects with dual hemispheric stimulation of the subthalamic nucleus (STN) and fornix/hypothalamus
Arm/Group | Deep Brain Stimulation
All-Cause Mortality (participants affected / at risk) | 1/5
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 3/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deep Brain Stimulation (N=5)
Seizure (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deep Brain Stimulation (N=5)
Sleep difficulty (Nervous system disorders) | 2 (2)
dystonia (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-15): https://cdn.clinicaltrials.gov/large-docs/41/NCT01563341/Prot_SAP_000.pdf